CLINICAL TRIAL: NCT00002251
Title: A Multiple Dose Crossover Pharmacokinetics Study to Evaluate the Effects of Food on the Absorption of Oral Ganciclovir
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 059A; ICM 1775
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1991-05

CONDITIONS: Cytomegalovirus Infections; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Ganciclovir; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome; Biological Availability
MeSH Terms: conditions — Cytomegalovirus Infections; HIV Infections; AIDS-Related Opportunistic Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Acquired Immunodeficiency Syndrome | interventions — Ganciclovir

INTERVENTIONS:
Drug: Ganciclovir

SUMMARY:
This study is designed to determine the influence of food on the absorption and relative bioavailability of oral ganciclovir by comparing the absorption of oral ganciclovir in a fed and fasting state at steady state plasma levels.

ELIGIBILITY:
Inclusion Criteria

Patients must have the following:

* Confirmation of HIV infection by HIV antibody testing, p24 antigen, or culture of HIV.
* Documented confirmation of present or past CMV infection.
* Must understand the nature of the study, agree to tests required in the protocol, and must understand and sign an informed Consent form approved by the appropriate Institutional Review Board and by Syntex.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Uncontrolled diarrhea or clinically significant gastrointestinal symptoms including persistent nausea or abdominal pain.

Concurrent Medication:

Excluded:

* Antimetabolites. Interferons. Other nucleoside analogs. Zidovudine (AZT). Any investigational drug.

Patients with the following are excluded:

* Any concomitant conditions listed in Exclusion Co-Existing Conditions.
* Karnofsky score < 70.
* Hypersensitivity to acyclovir.
* Displaying signs of dementia or decreased mentation which would interfere with the ability of the subject to follow protocol schedule.

Prior Medication:

Excluded:

* Anti-cytomegalovirus therapy including ganciclovir therapy for treatment of CMV disease.
* Excluded within 4 days of study entry:
* Antimetabolites.
* Interferons.
* Other nucleoside analogs.
* Zidovudine (AZT).

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Davies Med Ctr, San Francisco, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia

REFERENCES:
- [Background] Lavelle J, Follansbee S, Trapnell CB, Buhles WC, Griffy KG, Jung D, Dorr A, Connor J. Effect of food on the relative bioavailability of oral ganciclovir. J Clin Pharmacol. 1996 Mar;36(3):238-41. doi: 10.1002/j.1552-4604.1996.tb04193.x. PMID 8690817